CLINICAL TRIAL: NCT02680821
Title: Effect of Reconstruction of the Anterolateral Ligament (ALL) in Combination With Revision Anterior Cruciate Ligament (ACL) Surgery. A Clinical Randomized Trial
Brief Title: Reconstruction of the Anterolateral Ligament (ALL) With Revision Anterior Cruciate Ligament (ACL) Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Danish EC - 1107232415
Record Dates: First submitted 2016-02-08; First posted 2016-02-12 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Rupture of Anterior Cruciate Ligament; Anterolateral Ligament Reconstruction
Keywords: Laxity; Knee; Rupture; ALL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Rupture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isolated ACL-revision (Other): The standard operation with an isolated Anterior cruciate ligament.
  Interventions: Procedure: ACL revision (Anterior cruciate ligament )
- Combined ACL and ALL surgery (Other): An operation with an Anterior cruciate ligament combined with an anterolateral ligament.
  Interventions: Procedure: ALL reconstruction (Anterolateral ligament); Procedure: ACL revision (Anterior cruciate ligament )

INTERVENTIONS:
Procedure: ALL reconstruction (Anterolateral ligament)
  Arms: Combined ACL and ALL surgery
Procedure: ACL revision (Anterior cruciate ligament )

SUMMARY:
Patients with combined Anterolateral ligament (ALL) reconstruction- Anterior cruciate ligament (ACL) revision will have a better rotational knee stability and therefore better patient reported outcome measure (PROM) scores compared to patients, who have ACL revision surgery without ALL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ACL revision surgery indication

Exclusion Criteria:

* Patients with difficulties of understanding danish

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2024-09 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Difference in The Knee Numeric-Entity Evaluation Score (KNEES) | 12 months
  questionaire

SECONDARY OUTCOMES:
Difference in Knee injury and Osteoarthritis Outcome Score (KOOS) | 12 Months
  questionaire
Difference in KT-1000 | 12 Months
  Objective Knee stability
Difference in TEGNER functional score | 12 Months
  questionaire

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Tage-Hansens Gade 2b, Aarhus, Denmark